CLINICAL TRIAL: NCT04198415
Title: Post-Marketing All-Patient Drug Use Results Study for Venetoclax in Japanese Patients With Relapsed and Refractory Chronic Lymphocytic Leukemia (Including Small Lymphocytic Leukemia)
Brief Title: A Study of the Safety and Efficacy of Venetoclax in Japanese Participants With Relapsed and Refractory Chronic Lymphocytic Leukemia (Including Small Lymphocytic Leukemia)
Acronym: VENCLL regPMOS
Status: Completed | Type: Observational
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Other Study IDs: P19-830
Record Dates: First submitted 2019-12-12; First posted 2019-12-13 (Actual); Last update posted 2023-10-19 (Actual); Status verified 2023-10

CONDITIONS: Cancer; Chronic Lymphocytic Leukemia (CLL); Small Lymphocytic Leukemia (SLL)
Keywords: Cancer; Chronic Lymphocytic Leukemia (CLL); Small Lymphocytic Leukemia (SLL); Relapsed/Refractory; Venetoclax
MeSH Terms: conditions — Neoplasms; Leukemia, Lymphocytic, Chronic, B-Cell; Recurrence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Venetoclax Participants: Participants prescribed and treated with venetoclax.

SUMMARY:
This study will collect real-world safety and efficacy data from Japanese relapse/refractory chronic lymphocytic leukemia (CLL) and small lymphocytic leukemia (SLL) participants treated with venetoclax.

ELIGIBILITY:
Inclusion Criteria:

-Prescribed and treated with venetoclax

Exclusion Criteria:

None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All participants treated with venetoclax per the local label.
Sampling Method: Non-Probability Sample
Enrollment: 4 (Actual)
Dates: Start 2020-02-03 (Actual); Primary Completion 2022-10-21 (Actual); Study Completion 2022-10-21 (Actual)

PRIMARY OUTCOMES:
Number of Participants With Adverse Events | Approximately 37 weeks
  An adverse event (AE) is defined as any untoward medical occurrence in a patient or clinical investigation participant administered a pharmaceutical product which does not necessarily have a causal relationship with this treatment. The investigator assesses the relationship of each event to the use of study drug as either probably related, possibly related, probably not related or not related. A serious adverse event (SAE) is an event that results in death, is life-threatening, requires or prolongs hospitalization, results in a congenital anomaly, persistent or significant disability/incapacity or is an important medical event that, based on medical judgment, may jeopardize the participant and may require medical or surgical intervention to prevent any of the outcomes listed above. Treatment-emergent adverse events/treatment-emergent serious adverse events (TEAEs/TESAEs) are defined as any event that began or worsened in severity after the first dose of study drug.
Overall Incidence of Averse Drug Reactions (ADRs) of Tumor Lysis Syndrome (TLS), Bone Marrow Suppression, and Infections | Approximately 37 weeks
  Adverse drug reactions were defined as AEs of which a causal relationship with venetoclax could not be ruled out. Overall incidence of ADRs of special interest (TLS, bone marrow suppression, and infections) will be collected.
Incidence of Adverse Drug Reactions (ADR) | Approximately 37 weeks
  Adverse drug reactions were defined as AEs of which a causal relationship with venetoclax could not be ruled out. All grades of ADRs will be collected.
Incidence of TLS According to Physician Assessment | Approximately 37 weeks
  Incidence of TLS according to physician assessment.
Incidence of TLS According to Howard Criteria | Approximately 37 weeks
  Incidence of TLS according to Howard criteria which is a classification system of TLS. Laboratory results must show two or more unusual measurements within a 24-hour period.
Incidence of Bone Marrow Suppression | Approximately 37 weeks
  Incidence of bone marrow suppression including neutropenia (all grades) and febrile neutropenia.
Incidence of Infections | Approximately 37 weeks
  Incidence of infections.
Incidence of ADRs When Venetoclax is Used Concomitantly with CYP3A Inhibitors | Approximately 37 weeks
  Incidence of ADRs when venetoclax is used concomitantly with CYP3A inhibitors will be collected.
Number of Prophylactic Measures Used for TLS | Approximately 37 weeks
  Number and description of prophylactic measures used in real-world clinical practice for TLS will be collected.
Number of Monitoring Measures Used for TLS | Approximately 37 weeks
  Number and description of monitoring measures used in real-world clinical practice for TLS will be collected.
Number of Participants with Dose Modifications | Approximately 37 weeks
  Summary data will be collected for participants with dose modifications.
Number of Participants with Dose Interruptions | Approximately 37 weeks
  Summary data will be collected for participants with dose interruptions.
Number of Participants Who Discontinued Venetoclax | Approximately 37 weeks
  Summary data will be collected for participants who discontinued treatment with venetoclax.
Best Overall Response Rate (ORR) | Approximately 37 weeks
  Defined as complete response (CR), complete response with incomplete marrow recovery (CRi), partial response (PR), nodular partial response (nPR) according to physician assessment based on International Workshop on Chronic Lymphocytic Leukemia (iwCLL) 2018 guidelines and Japanese Society of Hematology clinical guidelines.
Time to Best Response | Approximately 37 weeks
  Time to best response according to physician assessment based on International Workshop on Chronic Lymphocytic Leukemia (iwCLL) 2018 guidelines and Japanese Society of Hematology clinical guidelines.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (102):
- Japan (102):
  - Japanese Red Cross Aichi Medical Center Nagoya Daini Hospital /ID# 239524, Nagoya, Aichi-ken
  - Nagoya University Hospital /ID# 225300, Nagoya, Aichi-ken
  - Nagoya City University Hospital /ID# 240820, Nagoya, Aichi-ken
  - Toyohashi Municipal Hospital /ID# 227433, Toyohashi, Aichi-ken
  - Akita University Hospital /ID# 228510, Akita, Akita
  - Chiba Aoba Municipal Hospital /ID# 224486, Chiba, Chiba
  - Kameda General Hospital /ID# 232142, Kamogawa-shi, Chiba
  - National Cancer Center Hospital East /ID# 225885, Kashiwa-shi, Chiba
  - Kimitsu Chuo Hospital /ID# 243748, Kisarazu-shi, Chiba
  - Japanese Red Cross Narita Hospital /ID# 230276, Narita-shi, Chiba
  - Juntendo University Urayasu Hospital /ID# 239735, Urayasu-shi, Chiba
  - Ehime University Hospital /ID# 229642, Toon-shi, Ehime
  - Fukuiken Saiseikai Hospital /ID# 239091, Fukui-shi, Fukui
  - Hamanomachi Hospital /ID# 224484, Fukuoka, Fukuoka
  - National Hospital Organization Kyushu Medical Center /ID# 244229, Fukuoka, Fukuoka
  - Kyushu University Hospital /ID# 231759, Fukuoka, Fukuoka
  - Fukuoka University Hospital /ID# 239750, Fukuoka, Fukuoka
  - Aso Iizuka Hospital /ID# 221140, Iizuka-shi, Fukuoka
  - Kitakyushu Municipal Medical Center /ID# 239525, Kitakyushu-shi, Fukuoka
  - Tokiwakai Jyoban Hospital /ID# 239752, Iwaki, Fukushima
  - Gifu Municipal Hospital /ID# 244231, Gifu, Gifu
  - Gifu University Hospital /ID# 225295, Gifu, Gifu
  - Ogaki Municipal Hospital /ID# 225886, Ogaki-shi, Gifu
  - Fujioka General Hospital /ID# 226840, Fujioka-shi, Gunma
  - Gunmaken Saiseikai Maebashi Hospital /ID# 225887, Maebashi, Gunma
  - Gunma Prefectural Cancer Center /ID# 231760, Ota-shi, Gunma
  - Hiroshima Red Cross Hospital & Atomic-bomb Survivors Hospital /ID# 230274, Hiroshima, Hiroshima
  - Kitami Red Cross Hospital /ID# 224190, Kitami-shi, Hokkaido
  - Steel Memorial Muroran Hospita /ID# 248003, Muroran-shi, Hokkaido
  - Sapporo Hokushin Hospital /ID# 221137, Sapporo, Hokkaido
  - Hokkaido University Hospital /ID# 227635, Sapporo, Hokkaido
  - Sunagawa City Medical Center /ID# 231761, Sunagawa, Hokkaido
  - Ako Central Hospital /ID# 230267, Ako-shi, Hyōgo
  - Hyogo Prefectural Amagasaki General Medical Center /ID# 221138, Amagasaki-shi, Hyōgo
  - Hyogo Medical University Hospital /ID# 224959, Nishinomiya-shi, Hyōgo
  - Hitachi General Hospital /ID# 218530, Hitachi-shi, Ibaraki
  - Ibaraki Prefectural Central Hospital /ID# 226745, Kasama-shi, Ibaraki
  - JA Toride Medical Center /ID# 248004, Toride-shi, Ibaraki
  - University of Tsukuba Hospital /ID# 229738, Tsukuba, Ibaraki
  - Ishikawa Prefectural Central Hospital /ID# 230275, Kanazawa, Ishikawa-ken
  - Iwate Prefectural Central Hospital /ID# 224191, Morioka, Iwate
  - Imakiire General Hospital /ID# 229643, Kagoshima, Kagoshima-ken
  - Imamura General Hospital /ID# 228512, Kagoshima, Kagoshima-ken
  - Imamura General Hospital /ID# 234007, Kagoshima, Kagoshima-ken
  - Medical Corporation Seijinkai Ikeda Hospital /ID# 248713, Kanoya-shi, Kagoshima-ken
  - Shonan Kamakura General Hospital /ID# 224958, Kamakura-shi, Kanagawa
  - Kawasaki Municipal Ida Hospital /ID# 226842, Kawasaki-shi, Kanagawa
  - Yokosuka Genrl Hospital Uwamachi /ID# 225294, Yokosuka-shi, Kanagawa
  - Kumamoto University Hospital /ID# 228511, Kumamoto, Kumamoto
  - Kumamoto Shinto General Hospital /ID# 224957, Kumamoto, Kumamoto
  - University Hospital Kyoto Prefectural University of Medicine /ID# 240577, Kyoto, Kyoto
  - JCHO Kyoto Kuramaguchi Medical /ID# 250196, Kyoto, Kyoto
  - Kyoto University Hospital /ID# 239090, Kyoto, Kyoto
  - Miyagi Cancer Center /ID# 227435, Natori-shi, Miyagi
  - Koga General Hospital /ID# 248005, Miyazaki, Miyazaki
  - Miyazaki Prefectural Nobeoka Hospital /ID# 248714, Nabeoka-shi, Miyazaki
  - Showa Inan General Hospital /ID# 227431, Komagane-shi, Nagano
  - National Hospital Organization Matsumoto Medical Center /ID# 224487, Matsumoto-shi, Nagano
  - Nagasaki University Hospital /ID# 223272, Nagasaki, Nagasaki
  - Nara Hospital Kinki University Faculty of Medicine, /ID# 224969, Ikoma-shi, Nara
  - Niigata University Medical & Dental Hospital /ID# 244227, Niigata, Niigata
  - Oita Prefectural Hospital /ID# 224967, Ōita, Oita Prefecture
  - Duplicate_Oita University Hospital /ID# 224118, Yufu-shi, Oita Prefecture
  - Okayama University Hospital /ID# 229641, Okayama, Okayama-ken
  - Okayama Medical Center /ID# 223271, Okayama, Okayama-ken
  - Naha City Hospital /ID# 227432, Naha, Okinawa
  - Shiroyama Hospital /ID# 225298, Habikino-shi, Osaka
  - Kansai Medical University Hospital /ID# 224956, Hirakata-shi, Osaka
  - Ikeda City Hospital /ID# 221139, Ikeda, Osaka
  - Osaka City General Hospital /ID# 224605, Osaka, Osaka
  - Daini Osaka Police Hospital /ID# 243746, Osaka, Osaka
  - Sakai City Medical Center /ID# 224970, Sakai-shi, Osaka
  - Minami Sakai Hospital /Id# 228513, Sakai-sh, Osaka
  - Saitama Medical University International Medical Center /ID# 232528, Hidaka-shi, Saitama
  - Japanese Red Cross Saitama Hospital /ID# 224966, Saitama-shi, Saitama
  - Shimane Prefectural Central Ho /ID# 227437, Izumo-shi, Shimane
  - Seirei Mikatahara General Hospital /ID# 225888, Hamamatsu, Shizuoka
  - Juntendo University Shizuoka Hospital /ID# 225297, Izunokuni-shi, Shizuoka
  - Shizuoka Saiseikai Genaral Hospital /ID# 238768, Shizuoka, Shizuoka
  - Shizuoka Cancer Center /ID# 239523, Sunto-gun, Shizuoka
  - Tokushima University Hospital /ID# 245090, Tokushima, Tokushima
  - Juntendo University Hospital /ID# 226744, Bunkyo-ku, Tokyo
  - Tokyo Medical And Dental University Hospital /ID# 226841, Bunkyo-ku, Tokyo
  - Tokyo Metropolitan Cancer and Infectious Diseases Center Komagome Hospital /ID# 224604, Bunkyo-ku, Tokyo
  - Tokyo Metropolitan Cancer and Infectious Diseases Center Komagome Hospital /ID# 240819, Bunkyo-ku, Tokyo
  - National Cancer Center Hospital /ID# 225296, Chuo-ku, Tokyo
  - Medical Plaza Edogawa /ID# 244232, Edogawa Ward, Tokyo
  - Edogawa Hospital /ID# 239386, Edogawa-ku, Tokyo
  - The Cancer Institute Hospital Of JFCR /ID# 224485, Koto-ku, Tokyo
  - Toranomon Hospital /ID# 224115, Minato-ku, Tokyo
  - The Jikei University Hospital /ID# 227434, Minato-ku, Tokyo
  - Japanese Red Cross Medical Center /ID# 225299, Shibuya-ku, Tokyo
  - NTT Medical Center Tokyo /ID# 224117, Shinagawa-ku, Tokyo
  - Japan Community Health care Organization Tokyo Yamate Medical Center /ID# 227436, Shinjuku-ku, Tokyo
  - Yamaguchi Grand Medical Center /ID# 224965, Hohu-shi, Yamaguchi
  - Fujisawa City Hospital /ID# 222585, Fujisawa-shi
  - Harasanshin Hospital /ID# 223309, Fukuoka
  - Hachinohe Red Cross Hospital /ID# 250953, Hachinohe-shi
  - Takenaka Medical Clinic /ID# 224964, Higashiomi-shi
  - Kawaguchi Municipal Medical Center /ID# 225301, Kawaguchi-shi
  - Okayama City General Medical Center /ID# 224116, Okayama
  - Yuri Kumiai General Hospital /ID# 248002, Yurihonjō

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Ito T, Kamimura T, Kiguchi T, Kato K, Takenaka R, Kobayashi M, Ito A, Sakai M, Izutsu K. Venetoclax treatment for chronic lymphocytic leukemia/small lymphocytic leukemia in Japan: post-marketing surveillance. Int J Hematol. 2024 Nov;120(5):613-620. doi: 10.1007/s12185-024-03832-x. Epub 2024 Aug 21. PMID 39167348
- See also: clinical study report synopsis — https://www.abbvieclinicaltrials.com/study/?id=P19-830#additional-resources-section